CLINICAL TRIAL: NCT02878512
Title: Comparative Evaluation of General Anesthesia (SEA) Using 0.5% Bupivacaine and Segmental Epidural Anesthesia (GA) for Percutaneous Nephro Lithotomy - A Retrospective Analysis
Brief Title: Segmental Epidural Anesthesia (SEA) V/S General Anesthesia for PCNL
Acronym: AnesthesiaPCNL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shakuntala Basantwani, Associate Professor, Maharashtra University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IEC/69/16
Record Dates: First submitted 2016-06-23; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Success Rate Under Segmental Epidural; Post Operative Pain
Keywords: Segmental Epidural; Regional Anesthesia for PCNL
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCNL under General Anesthesia (Active Comparator): Patients were premedicated with Inj. Atropine 0.06 mg intramuscularly half an hour prior to surgery, IV ranitidine 1mg kg-1, IV ondansetron 0.08mg kg-1 IV midazolam 0.02mg kg-1 and Pentazocine 0.3 mg/kg. Anaesthesia was induced with IV Thiopentone sodium 3-5 mg kg-1 and Vecuronium 0.1mg kg-1.and then intubated. Anaesthesia was maintained on 50 %:50% nitrous oxide and oxygen, vecuronium and propofol infusion . At the end of the surgery postoperative analgesia was given with IV tarmadol and local nfiltration with 0.25% bupivacaine at the surgical site. Patients were reversed with IV glycopyrrolate 0.008mg kg-1 and IV neostigmine 0.06mg kg-1 and extubated.
  Interventions: Procedure: PCNL under General Anesthesia
- PCNL under Segmental epidural Anesthesia (Experimental): epidural space was located at T12 -L1 or L1-L2 space .The epidural catheter was inserted cephalad 5 cm upwards in the epidural space (tip approximately at T8 to T9). and test dose of 3 ml of 2% Adrenalized Lignocaine was administered..loading dose of 0.5% Bupivacaine, approximately 8 to 10 ml was injected epidurally with regular negative aspiration to block T6- T12 segments, if desired level was not achieved then additional dose of 1 to 1.5 ml 0.5% bupivacaine per spared segment was given to achieve the desired level.Motor blockade of the lower limbs was checked and noted before lithotomy, before prone and at the end of the surgery using Bromage scale. After two segment regression of sensory level epidural top up with 1/4th of initial dose 2 to 3 ml of 0.5% Bupivacaine was given. At the end of the surgery 8ml of 0.125% Bupivacaine was administered for postoperative analgesia and the catheter was removed.
  Interventions: Procedure: Segmental Epidural Anesthesia

INTERVENTIONS:
Procedure: PCNL under General Anesthesia — Patients undergoing percutaneous Nephrolithotomy received General anesthesia.
  Arms: PCNL under General Anesthesia
Procedure: Segmental Epidural Anesthesia — Patients undergoing PCNL surgery received Segmental epidural anesthesia with 0.5% bupivacaine.
  Other Names: Regional Anesthesia
  Arms: PCNL under Segmental epidural Anesthesia

SUMMARY:
Management of nephrolithiasis has been revolutionized by the advent of shock-wave lithotripsy (ESWL) and percutaneous nephrolithotomy (PCNL). PCNL is a minimally invasive endoscopic technique and is used for the fragmentation and removal of stones of size more than 20 to 30 mm, staghorn stones or multiple stones resistant to ESWL. Anaesthesia for PCNL is a challenge because of the disease, surgical procedure, positioning, hypothermia,and the possibility of fluid absorption, dilutional anaemia and blood loss. General anaesthesia is the gold standard for this surgery.The advent of new drugs has refined the technique of general anaesthesia. However there are several issues related to prone position still to be addressed like accidental extubation and difficult reintubation, nerve injuries and post operative respiratory complications.

Combined spinal epidural(CSE) and only epidural anaesthesia (EA) is a well established technique of anaesthesia for upper abdomen and lower thoracic surgeries. It use has also been reported in PCNL surgeries.Segmental epidural can selectively blocks pain fibres from the surgical site. This not only allows to limit the dose of the local anaesthetics, but also limit motor and sympathetic blockade. Selective sympathetic block is associated with respiratory, cardiac, gastrointestinal and metabolic benefits. This formed the basis of our current study. In the present study the investigators aimed to evaluate the efficacy of segmental epidural for PCNL and compared it with standard technique i.e. GA.

DETAILED DESCRIPTION:
To evaluate efficacy the investigators compared intraoperative haemodynamics, surgical clearance of stones, post operative pain, surgeon's and Patient's satisfaction scores and postoperative complications and side effects in 60 ASA I and II patients undergoing PCNL surgery who received either General anesthesia or Segmental epidural Anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II
* Age - 18 years to 60 years
* Either sex
* BMI < 30

Exclusion Criteria:

* Unwilling for consent
* ASA 3
* Obesity with BMI > 30.
* Contraindications for Epidural Anaesthesia
* Undilated pelvicalyceal system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hemodynamic parameters: Change in heart rate per minute from baseline | Every 15 minutes for 2 hours and then every hourly till 24 hours
  Change in heart rate per minute from baseline
Postoperative Pain using VAS | Postoperatively every hourly for 24 hours
  Post operative pain was studied using VAS
Hemodynamic parameters; change in Mean arterial pressures in mm Hg from baseline | Hemodynamic parameters Change in Mean Arterial Pressure in mm Hg Every 15 minutes for 2 hours and then every hourly till 24 hours
  change in mean arterial pressure from baseline

SECONDARY OUTCOMES:
Surgeon satisfaction score | 10 minutes Postoperative
  (0-extremely poor, 1-poor, 2-fair, 3-good, 4-excellent).

IPD SHARING:
Plan to Share IPD: No